CLINICAL TRIAL: NCT02186587
Title: CT-navigated, Patient-specific Custom Total Knee Replacement Versus Standard Total Knee Replacement: Comparison With a Marker-less Gait Analysis System and Validated Outcome Scores
Brief Title: iTotal Pilot Study of ConforMIS Custom Total Knee Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1206872
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Knee Arthroplasty, Total

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ConforMIS (Other): Subjects who receive a ConforMIS custom total knee implant.
  Interventions: Device: ConforMIS custom total knee

INTERVENTIONS:
Device: ConforMIS custom total knee — Total knee arthroplasty using ConforMIS custom total knee system with follow-up at 6 months

SUMMARY:
To compare the outcomes of patients receiving the ConforMIS custom total knee implant to the outcomes of patients who receiving an off-the-shelf total knee implant.

Hypothesis: Patient-specific, custom total knee implants manufactured from patient CT data, and implanted with CT-navigated custom instruments will show faster functional recovery, including gait and patient functional outcome scores, when compared to standard, off-the-shelf total knee components inserted with non-navigated instruments (the present standard of care in total knee surgery).

DETAILED DESCRIPTION:
The experimental design was changed based on enrollment hurdles to be a single cohort observational study where ConforMIS patients were enrolled and followed for 6 months with 6 minute walk used as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

- undergoing total knee arthroplasty

Exclusion Criteria:

- BMI >40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonny Bal, MD, Principal Investigator — Professor - PI
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ConforMIS: Subjects in this arm will receive a ConforMIS custom total knee implant.
  ConforMIS custom total knee
- Off-the-shelf: Subjects in this arm will receive an off-the-shelf total knee implant.
  Off-the-shelf total knee implant
Period: Overall Study
Arm/Group | ConforMIS | Off-the-shelf
Started | 28 | 0
Completed | 23 | 0
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- ConforMIS: Subjects in this arm will be having a ConforMIS custom total knee implant as part of standard of care.
  ConforMIS custom total knee
- Off-the-shelf: Subjects in this arm will receive an off-the-shelf total knee implant as part of standard of care.
  Off-the-shelf total knee implant
- Total: Total of all reporting groups
Arm/Group | ConforMIS | Off-the-shelf | Total
Number analyzed (Participants) | 28 | 0 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 19 |  | 19
  >=65 years | 9 |  | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 |  | 18
  Male | 10 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Distance Measured During 6-minute Walk Test
Description: Subjects will walk for 6 minutes and the distance covered will be measured in feet.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | ConforMIS
Number analyzed (Participants) | 23
feet | 1060 (373)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ConforMIS | Off-the-shelf
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/0
Other Adverse Events (participants affected / at risk) | 1/28 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ConforMIS (N=28) | Off-the-shelf (N=0)
knee stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No